CLINICAL TRIAL: NCT02153320
Title: A Long-term Follow-up of a Phase I/II Study to Compare the Persistence and to Perform in Depth Characterisation of the Cellular and Humoral Immune Response Following Vaccinations With GSK Biologicals' Candidate Vaccines Containing HBsAg and Different Adjuvants in Healthy Adult Volunteers
Brief Title: Study to Evaluate the Persistence of the Cellular and Humoral Immune Response Following Vaccinations With GlaxoSmithKline (GSK) Biologicals' Candidate Vaccines Containing HBsAg and Different Adjuvants in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 105721
Record Dates: First submitted 2014-05-22; First posted 2014-06-03 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis B
Keywords: HBsAg; Persistence of the immune response; Adjuvants
MeSH Terms: conditions — Hepatitis B | interventions — Blood Specimen Collection

ARMS (3):
- HBsAg + adjuvant 1 Group (Experimental): Single blood sample taken from subjects who had received GSK candidate vaccine containing HBsAg together with an adjuvant 1 in study 287615 (NCT00508833).
  Interventions: Procedure: Blood Sampling
- HBsAg + adjuvant 2 Group (Experimental): Single blood sample taken from subjects who had received GSK candidate vaccine containing HBsAg together with an adjuvant 2 in study 287615 (NCT00508833).
  Interventions: Procedure: Blood Sampling
- HBsAg + adjuvant 3 Group (Experimental): Single blood sample taken from subjects who had received GSK candidate vaccines containing HBsAg together with an adjuvant 3 in study 287615 (NCT00508833).
  Interventions: Procedure: Blood Sampling

INTERVENTIONS:
Procedure: Blood Sampling — Single blood sample taken from subjects who had participated in the study 287615 (NCT00508833).

SUMMARY:
The purpose of this long-term follow-up study was to evaluate the persistence of the cellular and the humoral immune response 4 years after the first dose of GSK Biologicals' investigational vaccine formulations containing HBsAg (used as a model antigen) and an adjuvant.

DETAILED DESCRIPTION:
Subjects in this long-term follow-up study were recruited among those subjects who completed the study 287615 (NCT00508833) and who were enrolled in specific groups. All subjects were vaccinated in the study 287615 (NCT00508833) according to a 0, 1, 10 month schedule. No new subjects were enrolled and no vaccine was administered in this long-term follow-up study. There was a single visit at Year 4 at which blood samples for immunogenicity assays were taken.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Subjects who took part in and completed study 287615 (NCT00508833).
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the blood sampling, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within three months prior to the blood sampling.
* Administration of immunoglobulins within the three months preceding the blood sampling or planned administration during the study period.
* Pregnant or lactating female.
* Documented HIV-positive subject.

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2005-09-05 (Actual); Primary Completion 2005-10-28 (Actual); Study Completion 2005-10-28 (Actual)

PRIMARY OUTCOMES:
Frequency of CD4 and CD8 T cells expressing IFN-γ and/or TNF-α and/or IL-2 and/or CD40L upon short term in vitro stimulation with HbsAg derived peptides using cytokine flow cytometry. | Week 48.
  The blood samples at Week 48 were taken during the primary study 287615 (NCT00508833).
Frequency of CD4 and CD8 T cells expressing IFN-γ and/or TNF-α and/or IL-2 and/or CD40L upon short term in vitro stimulation with HbsAg derived peptides using cytokine flow cytometry. | Week 78.
  The blood samples at Week 78 were taken during the primary study 287615 (NCT00508833).
Frequency of CD4 and CD8 T cells expressing IFN-γ and/or TNF-α and/or IL-2 and/or CD40L upon short term in vitro stimulation with HbsAg derived peptides using cytokine flow cytometry. | Year 4.

SECONDARY OUTCOMES:
Anti-HBs antibody titres as measured by ELISA. | Week, 48, Week 78, Year 4.
  The blood samples at Week 48 and Week 78 were taken during the primary study 287615 (NCT00508833).
Exploratory analysis of proteins and low molecular weight biomolecules in the serum using ELISA and other techniques to be defined. | Day 0, Day 1.
  The blood samples at Day 0 and Day 1 were taken during the primary study 287615 (NCT00508833).
Frequency of HBsAg specific memory B cells by B Cell Elispot assay. | Week 48, Week 78, Year 4.
  The blood samples at Week 48 and Week 78 were taken during the primary study 287615 (NCT00508833).
Frequency of HBs-specific or non specific T regulatory cells using cytokine flow cytometry and other techniques to be defined. | Day 0, Week 6, Week 46, Week 48.
  The blood samples at Day 0, Week 6, Week 46 and Week 48 were taken during the primary study 287615 (NCT00508833).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent

REFERENCES:
- See also: Results for study 105721 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/105721?search=study&b%22b''%22#rs